CLINICAL TRIAL: NCT06011668
Title: THE EFFECT OF DISTRACTION METHODS ON PAIN AND ANXIETY DURING INTRAMUSCULAR INJECTION IN CHILDREN AGED 6-12 YEARS
Brief Title: EFFECT OF DISTRACTION METHODS ON PAIN AND ANXIETY DURING INTRAMUSCULAR INJECTION IN CHILDREN
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Senem Merve KURT, Principal Investigator, Mersin University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: SKURT-001
Record Dates: First submitted 2023-08-12; First posted 2023-08-25 (Actual); Last update posted 2023-08-25 (Actual); Status verified 2023-08

CONDITIONS: Pain, Acute; Anxiety and Fear
Keywords: Pain; Anxiety; Distraction; Children; Intramuscular injection
MeSH Terms: conditions — Acute Pain; Anxiety Disorders; Pain

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- distraction method (Experimental): video game playing
  Interventions: Device: video game playing, kaleidoscope and virtual reality glasses
- distraction (Experimental): kaleidoscope
  Interventions: Device: video game playing, kaleidoscope and virtual reality glasses
- distraction methods (Experimental): virtual reality glasses
  Interventions: Device: video game playing, kaleidoscope and virtual reality glasses

INTERVENTIONS:
Device: video game playing, kaleidoscope and virtual reality glasses — This thesis study was conducted with randomized controlled methods for control in order to analyze the effect of drawing attention to different directions during intramuscular use in countries to what extent the methods of drawing attention to pain and anxiety.

SUMMARY:
This thesis study was conducted in an unblinded, randomized controlled experimental manner in order to analyze the effect of attention-drawing methods that can be used during intramuscular injection in children on pain and anxiety.

DETAILED DESCRIPTION:
Data were collected in the Pediatric Emergency Injection Unit of Mersin City Training and Research Hospital between October and December 2021. Children aged 6-12 years were included in the study. In the study, the sample was divided into four groups. The study consisted of 180 children, 45 children in each group. Using the randomization program, it was determined which sample group the children would be included in.

In the study, video game playing, kaleidoscope and virtual reality glasses were used as a distraction method for the experimental group. Intramuscular injection (IM) was applied to the control group without any application. The research implementation period lasted an average of one minute. Required ethical permissions were obtained prior to the research. Wong-Baker Faces Pain Scale (WBFPRS) was used to measure pain level and Child Fear Scale (CFS) was used to measure anxiety level in the study. Explanatory information about the application to be made to the children and their parents was given by the researcher, and the consent form was signed by informing them voluntarily. The research data were collected by the researcher by interviewing the children face to face. In line with the data obtained in the study, it was concluded that the descriptive characteristics of the children in the experimental and control groups were similar (p>0.05). It was concluded that playing video games, kaleidoscope, and virtual reality glasses, among the distraction methods applied in the study, reduced pain and anxiety. It is expected that techniques that reduce pain and anxiety when intramuscular injections are given to children in nursing practices will be used in practice and that these practices will be included in the training of nurses.

ELIGIBILITY:
Inclusion Criteria:

* Children between the ages of 6-12 and their families who speak Turkish and accepted the voluntary informed consent form verbally and in writing.
* Children who do not have a chronic disease (Children with chronic diseases such as DM, asthma, hypertension, meningitis, epilepsy, etc. will not be included in the study as their response levels to pain will vary.)
* Children who have not taken an analgesic drug in the last 6 hours
* No physical or mental illness
* Children who have no suspicion of covid 19 transmission in their family or themselves
* Children whose vital signs are in parameters suitable for their age will be taken.

Exclusion Criteria:

* Children who did not accept the voluntary informed consent form verbally and in writing
* Children with chronic diseases (Children with chronic diseases such as DM, asthma, hypertension, meningitis, epilepsy, etc. will not be included in the study as their response levels to pain will vary.)
* Children who have taken an analgesic drug in the past 6 hours
* Those who have a suspected covid 19 transmission in their family or themselves
* Children with any physical or mental illness will not be included.

Ages: 6 Years to 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 180 (Actual)
Dates: Start 2021-10-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-12-15 (Actual)

PRIMARY OUTCOMES:
Pain was measured by Wong- Baker Faces Pain Scale | at 1st minute before the procedure
  The scale, which was developed by Wong and Baker in 1981 and renewed in 1983, is one of the most common methods used in pain assessment. The use of the scale is suitable for 3 years old and above. Before using the scale, the pain level of the statements on the scale should be explained to the child.
Pain was measured by Wong- Baker Faces Pain Scale | during the procedure
  The scale, which was developed by Wong and Baker in 1981 and renewed in 1983, is one of the most common methods used in pain assessment. The use of the scale is suitable for 3 years old and above. Before using the scale, the pain level of the statements on the scale should be explained to the child.
Pain was measured by Wong- Baker Faces Pain Scale | at 1st minute after the procedure
  The scale, which was developed by Wong and Baker in 1981 and renewed in 1983, is one of the most common methods used in pain assessment. The use of the scale is suitable for 3 years old and above. Before using the scale, the pain level of the statements on the scale should be explained to the child.
Fear was measured by Child Fear Scale | at 1st minute before the procedure
  In this scale, in which neutral anxiety expression is indicated as (0) and high level of anxiety/fear is indicated as (4), there are facial expressions that progress gradually from neutral anxiety expression to high level of anxiety.
Fear was measured by Child Fear Scale | during the procedure
  In this scale, in which neutral anxiety expression is indicated as (0) and high level of anxiety/fear is indicated as (4), there are facial expressions that progress gradually from neutral anxiety expression to high level of anxiety.
Fear was measured by Child Fear Scale | at 1st minute after the procedure
  In this scale, in which neutral anxiety expression is indicated as (0) and high level of anxiety/fear is indicated as (4), there are facial expressions that progress gradually from neutral anxiety expression to high level of anxiety.

CONTACTS AND LOCATIONS:
Locations (1):
- Senem Merve KURT, Mersin, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No